CLINICAL TRIAL: NCT04976634
Title: An Open-label, Multicenter, Phase 2 Study to Evaluate the Efficacy and Safety of Pembrolizumab Plus Lenvatinib in Combination With Belzutifan in Multiple Solid Tumors
Brief Title: Pembrolizumab Plus Lenvatinib in Combination With Belzutifan in Solid Tumors (MK-6482-016)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-016; MK-6482-016 (Other: MSD); 2023-503905-12-00 (EU CTIS Number); U1111-1288-3020 (Registry Identifier: UTN); 2020-005007-40 (EudraCT Number)
Record Dates: First submitted 2021-07-16; First posted 2021-07-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab; belzutifan; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Pembrolizumab + Belzutifan + Lenvatinib (Experimental): Participants will receive pembrolizumab 400 mg PLUS belzutifan 120 mg PLUS lenvatinib 20 mg (For HCC: 8 mg [body weight <60kg] or 12 mg [body weight ≥ 60 kg]). Pembrolizumab will be administered via intravenous (IV) infusion once every 6 weeks (Q6W) for a maximum of 18 doses (approximately 2 years). Belzutifan and lenvatinib will be administered orally once daily (QD) until progressive disease or discontinuation.
  Interventions: Drug: Pembrolizumab; Drug: Belzutifan; Drug: Lenvatinib
- Arm 2: Pembrolizumab + Lenvatinib (Experimental): Participants with IO resistant ESCC will receive pembrolizumab 400 mg PLUS lenvatinib 20 mg. Pembrolizumab will be administered via intravenous (IV) infusion once every 6 weeks (Q6W) for a maximum of 18 doses (approximately 2 years). Lenvatinib will be administered orally once daily (QD) until progressive disease or discontinuation.
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 400 mg administered Q6W via IV infusion
  Other Names: MK-3475; KEYTRUDA®
Drug: Belzutifan — Belzutifan 120 mg administered QD via oral tablet
  Other Names: MK-6482; PT2977; WELIREG™
  Arms: Arm 1: Pembrolizumab + Belzutifan + Lenvatinib
Drug: Lenvatinib — Lenvantinib dose for HCC is 8 mg QD for body weight <60 kg and 12 mg QD for body weight ≥ 60 kg administered via oral capsule. For all other tumors, the lenvatinib dose is 20 mg QD administered via oral capsule
  Other Names: MK-7902; E7080; LENVIMA®

SUMMARY:
The purpose of this study is to determine the safety and efficacy of belzutifan in combination with pembrolizumab and lenvatinib in multiple solid tumors including hepatocellular carcinoma (HCC), colorectal cancer (CRC), pancreatic ductal adenocarcinoma (PDAC), biliary tract cancer (BTC), endometrial cancer (EC),and esophageal squamous cell carcinoma (ESCC). There is no formal hypothesis testing in this study.

DETAILED DESCRIPTION:
Effective as of Amendment 3 (26 Mar 2025), enrollment of participants with ESCC will be closed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following advanced (unresectable and/or metastatic) solid tumors, documented by histopathology or cytopathology:

  * Hepatocellular carcinoma (HCC)
  * Colorectal cancer (CRC) (non-microsatellite instability-high [non-MSI-H]/deficient mismatch repair [dMMR])
  * Pancreatic ductal adenocarcinoma (PDAC).
  * Biliary tract cancer (BTC) (includes intrahepatic, extrahepatic cholangiocarcinoma [CCA] and gall bladder cancer)
  * Endometrial cancer (EC)
  * Esophageal squamous cell carcinoma (ESCC)
* Disease progression on or since the most recent treatment (does not apply to newly diagnosed unresectable or metastatic HCC or EC).
* Measurable disease per RECIST v1.1 as assessed locally (by investigator) and verified by BICR
* Submission of an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Male participants are abstinent from heterosexual intercourse or agree to follow contraceptive guidance during and for at least 7 days after last dose of study intervention with belzutifan and lenvatinib
* Female participants are not pregnant or breastfeeding, not a woman of child-bearing potential (WOCBP), or is a WOCBP and agrees to follow contraceptive guidance during the intervention period and and for at least 120 days after the last dose of pembrolizumab or for at least 30 days after last dose of lenvatinib or belzutifan, whichever occurs last
* Adequate organ function
* Adequately controlled blood pressure with or without antihypertensive medications
* HCC Specific Inclusion Criteria: No prior systemic chemotherapy, including anti-VEGF therapy, anti-programmed cell-death (PD-1)/PD-L1 or any systemic investigational anticancer agents for advanced/unresectable HCC (1L)
* CRC ([non-MSI-H/dMMR) Specific Inclusion Criteria: Received at least 2 prior lines of systemic therapy for unresectable or metastatic disease which includes fluoropyrimidine, irinotecan and oxaliplatin
* PDAC Specific Inclusion Criteria: Prior therapy with at least 1 (platinum or gemcitabine containing regimen) but no more than 2 prior systemic therapies for unresectable or metastatic pancreatic cancer
* BTC Specific Inclusion Criteria: Received at least 1 prior line of systemic therapy (containing gemcitabine or fluoropyrimidine) for unresectable or metastatic disease
* EC Specific Inclusion Criteria: Study treatment is for 1L therapy of EC and participants should not have received prior systemic chemotherapy. Exception: May have received 1 prior line of line of systemic platinum-based adjuvant and/or neoadjuvant chemotherapy in the setting of a curative-intent resection, if the recurrence occurred ≥6 months after the last dose of chemotherapy or may have received prior radiation with or without chemotherapy
* ESCC Specific Inclusion Criteria: Have experienced radiographic or clinical progression on one prior line of standard systemic therapy (immune oncology (IO) naïve participants) or an anti-PD-1/PD-L1 (IO resistant participants)

Exclusion Criteria:

* Unable to swallow orally administered medication or presence of a gastrointestinal (GI) disorder that may affect study intervention absorption
* History of a second malignancy that is progressing or has required active treatment within 3 years
* A pulse oximeter reading <92% at rest, or requirement of intermittent supplemental oxygen/ chronic supplemental oxygen
* Presence of central nervous system (CNS) metastases and/or carcinomatous meningitis
* Clinically significant cardiovascular disease within 6 months of first dose of study intervention
* Symptomatic pleural effusion, unless clinically stable after treatment
* Preexisting ≥ Grade 3 gastrointestinal (GI) or non-GI fistula
* Moderate to severe hepatic impairment
* Clinically significant history of bleeding within 3 months before screening
* Presence of serious active nonhealing wound/ulcer/bone fracture
* Requirement for hemodialysis or peritoneal dialysis
* History of human immunodeficiency virus (HIV) infection
* History of Hepatitis B or active Hepatis C virus infections. with exceptions for HCC and BTC
* Prior therapy with a PD-1, anti-PD-L1, anti-PD-L2 agent, vascular endothelial growth factor (VEGF) tyrosine kinase inhibitor (TKI) or hypoxia-inducible factor 2α (HIF-2α)
* Radiographic evidence of intratumoral cavitation, or invasion/infiltration of a major blood vessel
* EC specific exclusion criteria: History of carcinosarcoma, endometrial leiomyosarcoma or other high-grade sarcomas, or endometrial stromal sarcomas
* ESCC specific exclusion criteria: Has clinically apparent ascites or pleural effusion or experienced weight loss >20% over approximately 3 months before first dose of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2027-03-22 (Estimated); Study Completion 2027-03-22 (Estimated)

PRIMARY OUTCOMES:
Arm 1: Number of Participants Who Experience at Least One Dose-limiting Toxicity (DLT) | Up to approximately 21 days
  Occurrence of any of the following will be considered a DLT if possibly, probably, or definitely related to study treatment administration: Grade 4 nonhematologic toxicity; Grade 4 hematologic toxicity lasting >7 days; Grade 4 thrombocytopenia-any duration; Grade 3 thrombocytopenia if associated with clinically significant hemorrhage; Febrile neutropenia Grade 3 or Grade 4; Grade 3 nonhematologic toxicity lasting >5 days despite optimal supportive care; Grade 3 hypertension not controlled by antihypertensive medication(s); Grade 3 or Grade 4 nonhematologic laboratory abnormality (if medical intervention is required, or leads to hospitalization, or persists for >1 week) ; Elevated bilirubin if persists >4 weeks (for HCC and BTC participants only); Designated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) liver test abnormalities; Treatment-related toxicity resulting in participant discontinuation of study intervention during the DLT window; Grade 5 toxicity.
Arm 1: Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 67 months
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience one or more AEs will be presented.
Arm 1: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 67 months
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be presented separately for the safety lead-in phase (up to 21 days) and the main study.
Confirmed Objective Response Rate (ORR) Per Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 67 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by BICR will be presented.

SECONDARY OUTCOMES:
Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 67 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Disease Control Rate (DCR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 67 months
  DCR is defined as the percentage of participants who have a CR, PR, or Stable Disease (SD). Per RECIST 1.1, CR = disappearance of all target lesions, PR = ≥30% decrease in the sum of product diameters (SPD) of target lesions, compared to baseline SPD, and SD = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. The best overall response of CR, PR, or SD after ≥ 6 weeks will be assessed per RECIST 1.1 by BICR.
Progression-Free Survival (PFS) Per RECIST 1.1 as Assessed by BICR | Up to approximately 67 months
  PFS is defined as the time from first day of study intervention to the first documented PD or death due to any cause, whichever occurs first as assessed by RECIST 1.1. PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 67 months
  OS is defined as the time from the first day of study intervention to death due to any cause.
ORR Per Modified Response Criteria in Solid Tumors Version 1.1 (mRECIST 1.1) for Hepatocellular Carcinoma (HCC) as Assessed by BICR | Up to approximately 67 months
  ORR, per mRECIST 1.1, is defined as the percentage of participants with CR (disappearance of any intratumoral arterial enhancement in all target lesions) or PR (at least a 30% decrease in the sum of diameters of viable [contrast enhancement in the arterial phase] target lesions, taking as reference the baseline sum of diameters of target lesions) as assessed by BICR. For participants with HCC, mRECIST1.1 allows assessment of treatment-related tumor necrosis and assessment of viable tumor by assessment with arterial phase imaging. ORR as assessed by BICR will be presented.
DOR Per mRECIST 1.1 for HCC as Assessed by BICR | Up to approximately 67 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in sum of diameters of target lesions) per mRECIST 1.1, DOR is defined as time from first documented evidence of CR or PR until progressive disease (PD) or death. Per mRECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters (SOD) of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. The mRECIST 1.1 this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ. For participants with HCC, mRECIST1.1 allows assessment of treatment-related tumor necrosis and assessment of viable tumor by assessment with arterial phase imaging. DOR as assessed by BICR will be presented.
DCR Per mRECIST 1.1 for HCC as Assessed by BICR | Up to approximately 67 months
  DCR is defined, per mRECIST 1.1, as the percentage of participants who have a CR (Disappearance of all target lesions) or PR (At least a 30% decrease in the sum of diameters of target lesions) or Stable Disease (SD, Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD [At least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]). For participants with HCC, mRECIST1.1 allows assessment of treatment-related tumor necrosis and assessment of viable tumor by assessment with arterial phase imaging. The best overall response of CR, PR, or SD after ≥ 6 weeks per mRECIST 1.1 for HCC will be assessed by BICR.
PFS Per mRECIST 1.1 for HCC as Assessed by BICR | Up to approximately 67 months
  PFS, per mRECIST 1.1, is defined as the time from first dose of study treatment to the first documented PD or death due to any cause, whichever occurs first as assessed by mRECIST1.1 to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. Per mRECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. For participants with HCC, mRECIST1.1 allows assessment of treatment-related tumor necrosis and assessment of viable tumor by assessment with arterial phase imaging. PFS as assessed by BICR will be presented.
Arm 2: Number of Participants Who Experience an AE | Up to approximately 67 months
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE after administration of pembrolizumab plus lenvatinib will be presented.
Arm 2: Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 67 months
  An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment of pembrolizumab plus lenvatinib after an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (57):
- United States (16):
  - University of Arizona Cancer Center-University of Arizona Cancer Center - North Campus ( Site 5047), Tucson, Arizona
  - City of Hope Comprehensive Cancer Center ( Site 5002), Duarte, California
  - Cedars-Sinai Medical Center ( Site 5045), Los Angeles, California
  - UCSF Medical Center at Mission Bay ( Site 5021), San Francisco, California
  - Yale-New Haven Hospital-Yale Cancer Center ( Site 5013), New Haven, Connecticut
  - Sibley Memorial Hospital ( Site 5051), Washington D.C., District of Columbia
  - University of Florida College of Medicine ( Site 5015), Gainesville, Florida
  - Johns Hopkins Hospital-Sidney Kimmel Comprehensive Cancer Center - GI and Immunology ( Site 5048), Baltimore, Maryland
  - Brigitte Harris Cancer Pavilion ( Site 5055), Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center ( Site 5050), New York, New York
  - Duke Cancer Institute ( Site 5026), Durham, North Carolina
  - University of Texas MD Anderson Cancer Center-Gastrointestinal Medical Oncology ( Site 5049), Houston, Texas
  - Inova Schar Cancer Institute ( Site 5039), Fairfax, Virginia
  - Blue Ridge Cancer Care ( Site 5053), Roanoke, Virginia
  - Northwest Medical Specialties, PLLC ( Site 5025), Tacoma, Washington
  - University of Wisconsin Hospitals and Clinics ( Site 5037), Madison, Wisconsin
- Australia (4):
  - Gosford Hospital-Oncology Trials ( Site 4004), Gosford, New South Wales
  - Westmead Hospital-Department of Medical Oncology ( Site 4001), Westmead, New South Wales
  - Northern Hospital-Department of Medical Oncology ( Site 4003), Epping, Victoria
  - Cabrini Hospital - Malvern-Cabrini Institute ( Site 4000), Malvern, Victoria
- Belgium (5):
  - Antwerp University Hospital-Oncology ( Site 1002), Edegem, Antwerpen
  - Cliniques universitaires Saint-Luc-Medical Oncology ( Site 1001), Brussels, Bruxelles-Capitale, Region de
  - UZ Leuven ( Site 1000), Leuven, Vlaams-Brabant
  - AZ Delta vzw ( Site 1004), Roeselare, West-Vlaanderen
  - Université Catholique de Louvain-Namur - Centre Hospitalier -Oncology ( Site 1003), Namur
- Chile (5):
  - Clínica Puerto Montt ( Site 3110), Port Montt, Los Lagos Region
  - FALP-UIDO ( Site 3102), Santiago, Region M. de Santiago
  - Oncovida ( Site 3108), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 3100), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 3107), Temuco, Región de la Araucanía
- France (7):
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer ( Site 1103), Rennes, Brittany Region
  - CHU Besançon-Medical oncology ( Site 1101), Besançon, Doubs
  - CHU Brest Cavale Blanche ( Site 1107), Brest, Finistere
  - Institut Regional du Cancer Montpellier ( Site 1106), Montpellier, Herault
  - Centre Hospitalier Universitaire de Grenoble-Medical Oncology ( Site 1105), La Tronche, Isere
  - Sainte Catherine Institut du Cancer Avignon Provence ( Site 1108), Avignon, Vaucluse
  - Hôpital Beaujon-Oncologie Digestive ( Site 1104), Clichy, Île-de-France Region
- Israel (4):
  - Rambam Health Care Campus-Oncology ( Site 1300), Haifa
  - Hadassah Medical Center-Oncology ( Site 1303), Jerusalem
  - Sheba Medical Center-ONCOLOGY ( Site 1302), Ramat Gan
  - Sourasky Medical Center-Oncology ( Site 1301), Tel Aviv
- Netherlands (3):
  - Maastricht UMC+-Medical Oncology ( Site 1501), Maastricht, Limburg
  - Leids Universitair Medisch Centrum-Medical Oncology ( Site 1504), Leiden, South Holland
  - Universitair Medisch Centrum Utrecht-Medical Oncology ( Site 1503), Utrecht
- New Zealand (2):
  - Auckland City Hospital-Liver Research Unit ( Site 4201), Grafton, Auckland
  - Auckland City Hospital-Cancer & Blood Research ( Site 4200), Auckland
- South Korea (6):
  - Chonnam National University Hwasun Hospital-Hemato-Oncology ( Site 4105), Hwasun Gun, Jeonranamdo
  - Keimyung University Dongsan Hospital CRC room 1 ( Site 4104), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital-Internal Medicine ( Site 4103), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 4100), Seoul
  - Asan Medical Center-Department of Oncology ( Site 4101), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 4102), Seoul
- Spain (5):
  - Hospital Germans Trias i Pujol-Instituto Catalán de Oncología de Badalona ( Site 1806), Badalona, Barcelona
  - CHUS - Hospital Clinico Universitario-Servicio de Oncologia ( Site 1807), Santiago de Compostela, La Coruna
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON ( Site 1801), Madrid, Madrid, Comunidad de
  - Hospital Universitario Central de Asturias-Medical Oncology ( Site 1802), Oviedo, Principality of Asturias
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 1800), Barcelona

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Gebrael G, Sahu KK, Agarwal N, Maughan BL. Update on combined immunotherapy for the treatment of advanced renal cell carcinoma. Hum Vaccin Immunother. 2023 Dec 31;19(1):2193528. doi: 10.1080/21645515.2023.2193528. Epub 2023 Apr 16. PMID 37062953
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26231&tenant=MT_MSD_9011